CLINICAL TRIAL: NCT06567756
Title: A Multicenter, Prospective, Randomized Controlled Clinical Trial of the Effect of Conformal Sphincter-preservation Operation Versus Intersphincteric Resection on Postoperative Anal Function in Patients With Low Rectal Cancer
Brief Title: Conformal Sphincter-Preservation Operation Versus InterSphincteric Resection on Anal Function in Low Rectal Cancer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Changhai Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSVIS
Record Dates: First submitted 2024-01-02; First posted 2024-08-23 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-01

CONDITIONS: Rectum Cancer
Keywords: low rectum cancer; CSPO; ISR; anal function
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (experimental group): CSPO group (Experimental): The distal rectum is isolated to the entrance of the internal and external sphincter space, and then an oblique resection line is designed under direct vision according to the tumor site and shape, ensuring that the distal and lateral margins are not less than 1 cm, and preserving the contralateral dentate line and intestinal wall as much as possible, and completing the anastomosis manually or with instruments.
  Interventions: Procedure: CSPO
- Group B (control group): ISR group (Active Comparator): Partial, subtotal, or complete resection of the internal sphincter and/or a portion of the longitudinal rectal muscle, expansion of the distal rectal incision margin into the anal canal or to the anal verge, and completion of colorectal-anal anastomosis manually or instrumentally
  Interventions: Procedure: ISR

INTERVENTIONS:
Procedure: CSPO — The distal rectum is freed to the entrance of the internal and external sphincter space, and then an oblique resection line is designed under direct vision according to the tumor site and shape, ensuring that the distal and lateral margins are not less than 1 cm, and preserving the contralateral dentate line and the intestinal wall as much as possible, and the anastomosis is completed manually or with instruments.
  Arms: Group A (experimental group): CSPO group
Procedure: ISR — Partial, subtotal, or total excision of the internal sphincter and/or a portion of the longitudinal rectal muscle, expansion of the distal rectal excision margin into the anal canal or to the anal verge, and completion of the colo-anal anastomosis manually or instrumentally.
  Arms: Group B (control group): ISR group

SUMMARY:
In this clinical trial, the investigators compared anal function, genitourinary function, quality of life, perioperative safety, and oncological prognosis after CSPO for patients with low rectal cancer, using ISR as a control, to provide high-level evidence-based medical evidence for the choice of anorectal preservation surgical approaches for patients with low rectal cancer.

DETAILED DESCRIPTION:
The CSPO surgical approach is a series of targeted improvements designed primarily on the basis of analyzing the causes of poor postoperative function of the ISR, while building on research on the ultrastructure of the pelvic floor anal canal. For these reasons, the investigators designed the present study to compare anal function, quality of life, perioperative safety, and oncologic prognosis after CSPO for patients with low rectal cancer, using ISR surgery as a control, and to provide high-level evidence-based medical evidence for the choice of anorectal preservation surgical modalities for patients with low rectal cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-75 years;
2. Pathologically confirmed: moderately & well-differentiated rectal cancer;
3. Low rectal cancer: lower edge of tumor ≦5cm from anal verge or ≦2cm from dentate line;
4. Tumor diameter: ≤3cm or <1/3 bowel circumference;
5. Tumor infiltration depth: cT1-2, Bordeaux/Rullier classification: type II-III;
6. Locally progressive rectal cancer (cT1-4N0-2M0): significant tumor downstaging and downgrading after preoperative neoadjuvant therapy, meeting the above criteria;
7. ASA score: I-III and ECOG score: 0-1;
8. Undergo elective TME for colorectal or colorectal-anal canal anastomosis;
9. Normal preoperative anal function: Wexner score <10, LARS score <20;
10. Agree to participate in the clinical trial and sign an informed consent form.

Exclusion Criteria:

1. Combination of synchronous or metachronous (within 5 years) malignant tumors;
2. Combined distant metastasis of the tumor;
3. Combined intestinal obstruction, intestinal perforation, or intestinal bleeding requiring emergency surgery;
4. Combined psychiatric disorders that do not allow them to understand and participate in the study;
5. Combined systemic diseases that cannot tolerate surgery;
6. Women who are pregnant or breastfeeding;
7. Other reasons, judged by the investigator, for not being suitable for participation in this clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2030-09 (Estimated)

PRIMARY OUTCOMES:
Wexner incontinence score | 12 months after protective stoma closure
  The scale was totaled from 0 to 20, with higher scores indicating more severe disease and poorer anal function.

SECONDARY OUTCOMES:
LARS scoreIncontinence Score | 12 months after protective stoma closure
  The total score of the scale was 0-42, the higher the score, the more severe the condition and the worse the anal function, 0-20 indicated no LARS, 21-29 indicated minor LARS, and 30-42 indicated major LARS.
Quality of Life Questionaire-Core 30 | 12 months after radical resection of rectal cancer and protective stoma closure
  A core scale for all cancer patients with 30 entries, each on a 4-point scale, rated 1 to 4. It can be categorized into 15 domains, with 5 functional domains (somatic, role, cognitive, emotional, and social functioning), 3 symptomatic domains (fatigue, pain, and nausea and vomiting), 1 domain of general health status/quality of life, and 6 single entries (each as a domain). The scores of the entries included in each domain were summed and divided by the number of entries included to obtain a score for that domain (Raw Score RS). In order to make the scores of each domain comparable with each other, a linear transformation was further performed using a polarization method to convert the rough score into a standardized score (SS) with values ranging from 0 to 100. Higher scores for the functional and general health domains indicate better functional status and quality of life, while higher scores for the symptom domain indicate more symptoms or problems (poorer quality of life).
Overall survival | 3 years
  Overall Survival (OS) is the time from the start of randomization to death from any cause, and it is one of the best efficacy endpoints in oncology clinical trials. OS is usually the preferred endpoint when patient survival can be adequately assessed.
Clavien-Dindo complication grading | perioperative period
  Grade 1 included minor risk events not requiring therapy (with exceptions of analgesic, antipyretic, antiemetic, and antidiarrheal drugs or drugs required for lower urinary tract infection). Grade 2 complications were defined as potentially life-threatening complications with the need of intervention or a hospital stay longer than twice the median hospitalization for the same procedure. Grade 2 was divided into 2 subgroups based on the invasiveness of the therapy selected to treat the complication; grade 2a complications required medications only and grade 2b an invasive procedure. Grade 3 complications were defined as complications leading to lasting disability or organ resection, and finally, a Grade 4 complication indicated death of a patient due to a complication.

IPD SHARING:
Plan to Share IPD: No